CLINICAL TRIAL: NCT05803681
Title: Capacitively Coupled Electric Fields in the Treatment of Acute Vertebral Fragility Fractures
Brief Title: CCEF in the Treatment of Acute VFFs: Randomized Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bari Aldo Moro (Other)
Collaborators: IGEA (Industry)
Responsible Party: Principal Investigator, Davide Bizzoca, MD, PhDs. PhDs in Public health, Clinical Medicine and Oncology. DiMePre-J, University of Bari, University of Bari Aldo Moro
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CCEFVBME
Record Dates: First submitted 2023-03-11; First posted 2023-04-07 (Actual); Last update posted 2023-04-07 (Actual); Status verified 2023-03

CONDITIONS: Vertebral Fracture; Osteoporotic Fractures
Keywords: acute vertebral fracture; vertebral fragility fracture; vertebral bone marrow edema;; osteoporosis; osteopenia; fragility fractures; biophysical stimulation; capacitive coupled electric fields (CCEF); MRI; spine; back pain; aging
MeSH Terms: conditions — Spinal Fractures; Osteoporotic Fractures; Osteoporosis; Bone Diseases, Metabolic; Back Pain

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- CCEF group (Experimental): In the CCEF Group, patients received, as an adjunct to the clinical study protocol, CCEF stimulation (Osteospine®, IGEA SpA, Carpi, Italy) 8 h/die for sixty days.
  Clinical study protocol: (1) bed rest for the first twenty-five days and subsequent mobilization with a three-point hyperextension brace; (2) antiresorptive therapy (75 mg risedronate tablet weekly); (3) supplemental calcium carbonate with 1000 mg of elemental calcium daily if needed based on serum calcium concentration; (4) Vitamin D (≤500 IU daily) if the serum 25-hydroxyvitamin D concentration at the time of screening was below 16 ng/ml). Analgesic therapy with paracetamol 1000mg tablets was assumed for seven days and further depending on pain intensity; patients were required to report on a specific sheet paracetamol assumption.
  Interventions: Device: Capacitive Coupled Electric Fields (CCEF)
- Control Group (Other): (1) bed rest for the first twenty-five days and subsequent mobilization with a three-point hyperextension brace; (2) antiresorptive therapy (75 mg risedronate tablet weekly); (3) supplemental calcium carbonate with 1000 mg of elemental calcium daily if needed based on serum calcium concentration; (4) Vitamin D (≤500 IU daily) if the serum 25-hydroxyvitamin D concentration at the time of screening was below 16 ng/ml). Analgesic therapy with paracetamol 1000mg tablets was assumed for seven days and further depending on pain intensity; patients were required to report on a specific sheet paracetamol assumption.
  Interventions: Other: Calssic clinical protocol

INTERVENTIONS:
Device: Capacitive Coupled Electric Fields (CCEF) — In the CCEF Group, patients received, as an adjunct to the clinical study protocol, CCEF stimulation (Osteospine®, IGEA SpA, Carpi, Italy) 8 h/die for sixty days.
  Arms: CCEF group
Other: Calssic clinical protocol — (1) bed rest for the first twenty-five days and subsequent mobilization with a three-point hyperextension brace; (2) antiresorptive therapy (75 mg risedronate tablet weekly); (3) supplemental calcium carbonate with 1000 mg of elemental calcium daily if needed based on serum calcium concentration; (4) Vitamin D (≤500 IU daily) if the serum 25-hydroxyvitamin D concentration at the time of screening was below 16 ng/ml). Analgesic therapy with paracetamol 1000mg tablets was assumed for seven days and further depending on pain intensity; patients were required to report on a specific sheet paracetamol assumption.
  Arms: Control Group

SUMMARY:
in recent years the search for therapeutic protocols that could enhance the VFFs healing, thus reducing bed rest-related complications and improving the quality of life of osteoporotic patients. In this context, biophysical stimulation with Capacitively Coupling Electric Fields (CCEF) together, antiresorptive therapy, vitamin D supplementation, and analgesic drugs could play a central role.

CCEF is a non-invasive type of biophysical stimulation used to enhance fracture repair and spinal fusion. Positive effects of CCEF have been reported in osteoporotic vertebral fractures to resolve chronic pain and in postoperative pain, disability, and quality of life after spinal fusion In a preliminary observational study, Piazzolla et al. showed a significantly faster VBME resolution and back pain improvement in patients suffering from VFFs.

DETAILED DESCRIPTION:
Between January 2015 and December 2020, patients referring to the spine centres participating in this multicentre randomized controlled trial with acute VFFs type OF1 or OF2 were included in the present study. Ethical clearance was obtained from our centre's clinical research ethics, as per the 1964 Declaration of Helsinki, and all patients gave informed consent before enrolment in the study.

ELIGIBILITY:
Inclusion Criteria:

* male and female;
* years≥ 60 years old;
* BMI ≤ 35 kg/cm2;
* fracture site between T10 and L3;
* pain at the VCF level;
* low back pain onset within twenty days;
* VBME>60% in MRI at baseline;
* VBME in a maximum of two vertebral bodies.

Exclusion Criteria:

* posterior wall /pedicle injury;
* previous vertebroplasty/ kyphoplasty;
* history of spine infection or tuberculosis;
* history of malignant tumours that could spread to the spine;
* concomitant rheumatoid arthritis or spondylarthritis;
* scoliosis ≥ 40° according to Cobb;
* thoracolumbar kyphosis>20° or thoracic kyphosis>70°;
* any contraindication to MRI;
* use of biomedical devices.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2020-11-30 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
VBME resolution in MRI | Changes of VMBE at 60 days FU
  MRI of the spine

SECONDARY OUTCOMES:
Pain improvement | Changes of pain at 180 days FU compared to baseline
  VAS
quality of life and back pain improvement | Improvement of quality of life at 180 days FU compared to baseline
  ODI (Oswestry Disability Index)

CONTACTS AND LOCATIONS:
Overall Officials: Davide Bizzoca, MD, PhDs, Principal Investigator — AOU Policlinico di Bari

REFERENCES:
- [Derived] Piazzolla A, Bizzoca D, Barbanti-Brodano G, Formica M, Pietrogrande L, Tarantino U, Setti S, Moretti B, Solarino G. Capacitive biophysical stimulation improves the healing of vertebral fragility fractures: a prospective multicentre randomized controlled trial. J Orthop Traumatol. 2024 Apr 15;25(1):17. doi: 10.1186/s10195-024-00758-2. PMID 38622334